CLINICAL TRIAL: NCT06430554
Title: Personalized Ventilatory Strategy Based on Ventilation-perfusion Mismatch and Lung Recruitability in Moderate-to-severe ARDS Patients
Brief Title: Personalized Ventilation Based on Ventilation-perfusion Mismatch and Lung Recruitability
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Fengmei Guo, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Zhongda Hospital, Southeast University, China, Zhongda Hospital
Other Study IDs: 2024ZDSYLL044-P01
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Distress Syndrome; Positive-Pressure Respiration; Mechanical Ventilation
Keywords: Acute respiratory distress syndrome;Positive end expiratory pressure; Prone Position; Ventilation/perfusion matching.
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will explore the effects of PEEP and position on regional lung ventilation-perfusion mismatch by electrical impedance tomography (EIT) in moderate-to-severe ARDS patients with different lung recruitability.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is characterized by impaired ventilation-perfusion matching, which not only indicates the severity of the condition but also contributes to ventilation-induced lung injury. Higher positive end-expiratory pressure (PEEP) and prone position could improve ventilation-perfusion mismatch by recruiting collapsed lungs and facilitating more homogeneous ventilation, but these benefits might depend on lung recruitability. The present study aims to elucidate the regional effect of PEEP(low and high) and body position(supine and prone) on the ventilation-perfusion matching. Also endeavors to establish correlations between alterations in ventilation-perfusion matching patterns and the inherent lung recruitability.

Participants will be deeply sedated and paralyzed, ventilated in volume-controlled with protective ventilation (tidal volume=6-8 mL/Kg of predicted body weight and respiratory rate set to obtain normal pH). Then the patients will be sequentially assigned to each of four conditions as follows:

Low PEEP, supine position; High PEEP, supine position; Low PEEP, prone position; High PEEP, prone position. High PEEP and low PEEP is defined as 15 cmH2O and 5 cmH2O (or airway opening pressure, either of which was higher) respectively. Each measurement (e.g., arterial blood gas analysis, respiratory parameters, hemodynamics, EIT measurements) will be performed at least 15 minutes after changing ventilator settings and at least 1 hour after changing body positions. The timing of turning patients from supine to prone position is determined by the clinical team.

To assess lung recruitability, a single-breath derecruitment maneuver will be performed by changing PEEP 15 to 5 cmH2O (or airway opening pressure, either of which was higher) in supine position. Patients with recruitment-inflation ratio over the median value are defined as high recruiters.

EIT data will be collected by standard device (Infinity C500, Drager, Germany) with a sample rate of 50 Hz. The EIT belt will be placed directly below the armpits, between the third and fifth intercostal spaces. This positioning of the EIT belt will be maintained consistently during both supine and prone positions. A bolus of 10 ml 5% NaCl will be injected during a respiratory pause (≥8 s) through the central venous catheter to assess lung ventilation and perfusion distributions. The primary endpoint is EIT-based ventilation-perfusion matching (V/Q match%).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. Moderate-to-severe ARDS as per the 2023 ESICM definition
3. Undergoing invasive mechanical ventilation
4. Planned prone position based on the attending physicians' decisions
5. Signed informed consent

Exclusion Criteria:

1. age ≥85 years
2. Pregnancy
3. Severe hemodynamic instability (> 30% increase in vasopressors in the last 6 hours or norepinephrine > 0.5 µg/kg/min)
4. Clinically suspected elevated intracranial pressure (>18 mm Hg)
5. Bronchopleural fistula
6. Contraindication to EIT monitoring (e.g. burns, pacemaker, thoracic wounds limiting electrode belt placement)
7. Severe hypernatremia (>170mmol/L)
8. Re-admission of patients already enrolled in this study, or patients who are participating in other studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated mechanically ventilated ARDS patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ventilation-perfusion matching (V/Q match%) | Through study completion (within 24 hours)
  corresponding to the pixels that are both ventilated and perfused divided by the total number of pixels ventilated and/or perfused

SECONDARY OUTCOMES:
percentage of dead space | Through study completion (within 24 hours)
  corresponding to the ventilated but nonperfused pixels divided by the total number of pixels ventilated and/or perfused
percentage of shunt | Through study completion (within 24 hours)
  corresponding to the perfused but nonventilated pixels divided by the total number of pixels ventilated and/or perfused
Respiratory system compliance | Through study completion (within 24 hours)
  The compliance of respiratory system
PaO2/FiO2 ratio | Through study completion (within 24 hours)
  PaO2/FiO2 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Fengmei Guo, PhD, MD, Study Chair — Nanjing Zhongda Hospital, Southeast University
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No